CLINICAL TRIAL: NCT05814848
Title: A Single-arm Prospective Study of Secondary Infusion of Relmacabtagene Autoleucel Injection for Relapsed or Refractory B-cell Lymphoma
Brief Title: A Study of Secondary Infusion of Relmacabtagene Autoleucel Injection for Relapsed or Refractory B-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029019
Record Dates: First submitted 2023-03-16; First posted 2023-04-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-03

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): For patients who had undergone at least one disease assessment after the first treatment of Relmacabtagene Autoleucel injection and whose disease status was not complete remission, the investigators decided to give the patients a second treatment of Relmacabtagene Autoleucel injection based on clinical practice, and the specific dosage was determined by the investigators according to the patient's condition and dose reserve.
  Interventions: Drug: Relmacabtagene Autoleucel Injection

INTERVENTIONS:
Drug: Relmacabtagene Autoleucel Injection — For patients who had undergone at least one disease assessment after the first treatment of Relmacabtagene Autoleucel injection and whose disease status was not complete remission, the investigators decided to give the patients a second treatment of Relmacabtagene Autoleucel injection based on clinical practice, and the specific dosage was determined by the investigators according to the patient's condition and dose reserve.
  Other Names: CARTEYVA

SUMMARY:
To evaluate the efficacy and safety of post-marketing Regiorense injection secondary infusion in the treatment of adult patients with relapsed or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
CD19-targeted chimeric antigen receptor T-cell therapy has shown remarkable efficacy in relapsed or refractory B-cell malignancies. However, CD19 CAR-T cells are still unable to induce durable remissions in some patients. Further therapeutic strategies remain to be explored for patients who fail to achieve complete remission (CR) or who relapse after CAR-T treatment. the mechanisms underlying the failure of CAR-T cell therapy may be diverse and not yet fully understood. It may be due to the patient's own poor T-cell function, immunosuppressive tumour microenvironment, loss of tumour-targeting antigen expression with antitumour therapy, and compromised CAR-T renewal in vivo, or T-cell depletion due to the tumour microenvironment. It has recently been demonstrated that CAR-T cells become functionally depleted, or CAR lost, with sustained exposure to tumour antigen stimulation (Good, C, 2021). Extensive clinical experience suggests that CAR-T cell expansion and persistence are required to achieve a durable response. In patients requiring follow-up therapy after failure of the first CAR-T cell infusion (CART1), one option is a second infusion of CD19 CAR-T cells (CART2) for retreatment, and a second infusion of CD19 CAR-T cells (CART2) is considered a possible approach to improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) was obtained from the patients.
* Diagnosed relapsed or refractory B-cell lymphomas

  1. diffuse large B-cell lymphoma-not otherwise specified
  2. diffuse large B-cell lymphoma transformed from follicular lymphoma
  3. grade 3b follicular lymphoma
  4. primary mediastinal large B-cell lymphoma
  5. high-grade B-cell lymphoma with MYC and BCL-2 and/or BCL-6 rearrangements (double/triple hit lymphoma)
  6. adult follicular lymphoma refractory to second-line or later systemic therapy or relapsed within 24 months Adult patients who had completed the first treatment with remifentanil injection;
* The patient had undergone at least one post-treatment disease assessment with Relmacabtagene Autoleucel Injection, and the investigator decided to retreat the patient (including PR\PD\SD) with commercially available Relmacabtagene Autoleucel injection based on clinical practice;
* Prior to the second infusion, an adequate dose of the manufactured product (80-150x106 CAR-T cells recommended) should be confirmed, at the investigator's discretion based on the patient's condition and dose stockpile；
* Confirmation of residual tumor tissue CD19+ in patients, if clinically permissible；
* Absence of antidrug antibody (ADA) to ricciolenz in plasma before retreatment；
* Toxicity associated with lymphocyte-clearing chemotherapy (fludarabine and cyclophosphamide), with the exception of alopecia, that resolved to ≤ grade 1 or returned to pre-first treatment levels before retreatment.
* The patients did not have serious adverse reactions during the first treatment, or the adverse reactions during the first treatment had resolved to the baseline level of the first treatment.

Exclusion Criteria:

* Patients with hypersensitivity to the active ingredient or any excipients (dimethyl sulfoxide, compound electrolyte injection, human serum albumin);
* Patients had uncontrolled systemic fungal, bacterial, viral, or other infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | three months
  Objective Response Rate (ORR) : The investigator-assessed best disease status of patients with relapsed or refractory B-cell lymphoma was the rate of Complete Response (CR) or Partial Response (PR) at 3 months after a second infusion of remifolenafil.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: No